CLINICAL TRIAL: NCT07261540
Title: Bilateral Knee Strength Asymmetry and Functional Performance in Older Women With Osteoarthritis
Acronym: STASFP-OA
Status: Completed | Type: Observational
Sponsor: Kocaeli Sağlık ve Teknoloji Üniversitesi (Other)
Responsible Party: Principal Investigator, Sena Çınarlı, Asisstant Professor, Kocaeli Sağlık ve Teknoloji Üniversitesi
Other Study IDs: KOSTU-25-OA-02
Record Dates: First submitted 2025-11-22; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-05

CONDITIONS: Knee Osteoarthristis; Postmenopausal Women; Functional Performance; Isokinetic Test; Muscle Strenght
Keywords: knee osteoarthristis; Postmenopausal women; muscle strenght; isokinetic test; Functional Performance
MeSH Terms: interventions — Walking Speed

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: Patients with bilateral knee osteoarthritis who met the inclusion criteria underwent a single laboratory assessment involving isokinetic strength testing, pain evaluation, dynamic balance assessment, and functional mobility tests. Isokinetic strength testing was performed on both knees of the patients.All assessments took 1 hour in total for each patient.
  Interventions: Other: Isokinetic Strength Testing

INTERVENTIONS:
Other: Isokinetic Strength Testing — Bilateral knee strength asymmetry was assessed using a Biodex System 4 Pro isokinetic dynamometer (Biodex Medical Systems, USA). Participants were securely positioned, and knee extensor and flexor strength were measured at angular velocities of 120°/s and 180°/s. Each participant performed five maximal concentric contractions per limb, with the highest peak torque values recorded.
  Other Names: Pain Assessment; Dynamic Balance Measurement; Functional Mobility; Gait Speed

SUMMARY:
Osteoarthritis (OA) is a degenerative joint disease that primarily affects the knees and becomes more prevalent with age. In individuals over 50, particularly those with bilateral knee osteoarthritis, it leads to chronic pain, limited mobility, and functional decline. This condition worsens due to muscle strength imbalances, especially in the quadriceps and hamstrings. These imbalances are triggered by pain, joint instability, and cartilage damage, which negatively impact muscle strength and coordination. In women, these asymmetries are more pronounced, increasing the risk of functional decline.

Recent studies highlight the significant role of strength asymmetry in functional limitations, affecting balance, gait, and daily activities. This study aims to investigate the impact of bilateral quadriceps and hamstring strength asymmetries on dynamic balance, gait efficiency, and functional mobility in older women with bilateral knee osteoarthritis.

The study aims to examine the effects of bilateral strength asymmetries in the knee extensors and flexors on dynamic balance, gait efficiency, and overall mobility in older women with bilateral knee osteoarthritis. We hypothesize that greater strength asymmetry will be associated with impaired dynamic balance, reduced gait efficiency, and decreased functional mobility.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a degenerative joint disease that commonly affects the knee, especially in individuals over 50. It leads to pain, reduced mobility, and functional decline. In bilateral knee OA, muscle imbalances, especially in the quadriceps and hamstrings, worsen functional limitations and increase the risk of falls. These imbalances are caused by pain, joint instability, and cartilage damage, affecting muscle strength and coordination. In older women, these issues are more pronounced, increasing their risk of functional decline compared to men.

Emerging research highlights the role of muscle strength asymmetry (differences between the left and right leg) in functional difficulties, such as poor balance, walking issues, and difficulty with daily tasks. This study aims to explore how these muscle imbalances in knee extensors and flexors impact overall functional abilities, such as balance and walking efficiency in women with bilateral knee OA.

The study seeks to examine how bilateral strength asymmetry in the knee muscles affects dynamic balance, gait efficiency, and mobility in older women with knee osteoarthritis. The hypothesis is that greater muscle imbalance will lead to worse balance, slower walking, and reduced mobility.

ELIGIBILITY:
Inclusion Criteria:

* women gender
* aged 50 years or older
* diagnosed with bilateral knee osteoarthritis (Kellgren-Lawrence grade II-III),
* capable of independent walking without assistive devices.

Exclusion Criteria:

* severe knee osteoarthritis requiring total knee arthroplasty
* neurological conditions affecting gait or balance
* severe musculoskeletal disorders
* uncontrolled systemic diseases
* cognitive impairments (Mini-Mental State Examination < 24)

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This cross-sectional observational study investigates the impact of bilateral isokinetic strength asymmetry on dynamic balance and gait speed in women with bilateral knee osteoarthritis. Participants were recruited from Inonu University Faculty of Medicine Research Hospital Physical Therapy and Rehabilitation Department with eligibility determined based on clinical and radiographic assessments.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-05-05 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Isokinetic Strength Testing | From enrollment to the end of evaluation in 1 hour
  Bilateral knee strength asymmetry was assessed using a Biodex System 4 Pro isokinetic dynamometer (Biodex Medical Systems, USA). Participants were securely positioned, and knee extensor and flexor strength were measured at angular velocities of 120°/s and 180°/s. Each participant performed five maximal concentric contractions per limb, with the highest peak torque values recorded. Higher asymmetry values indicated greater strength imbalances between limbs
Functional Mobility | From enrollment to the end of evaluation in 1 hour
  The 30-second Sit-to-Stand test was used to assess lower limb functional strength and endurance. Participants were instructed to stand up and sit down as many times as possible in 30 seconds from a standard chair (seat height: 46 cm) without using their arms. The total number of completed repetitions was recorded. A lower Sit-to-Stand score indicates reduced quadriceps endurance, decreased functional independence, and a higher fall risk in older adults.

SECONDARY OUTCOMES:
Pain Assessment | From enrollment to the end of evaluation in 1 hour
  Knee pain intensity during daily activities and strength testing was evaluated using the 10-cm Visual Analog Scale, a widely validated tool for assessing subjective pain perception in bilateral knee osteoarthritis patients
Dynamic Balance Measurement | From enrollment to the end of evaluation in 1 hour
  Dynamic balance was assessed using the Biodex Balance System (Biodex Medical Systems, Shirley, NY, USA), a validated system for evaluating postural control and stability. Participants performed the Limits of Stability (LOS) test, which measures movement control in eight directions, quantifying reaction time, movement velocity, endpoint excursion, and directional control
Gait Speed | From enrollment to the end of evaluation in 1 hour
  Gait speed was assessed using a 4-meter walk test, a reliable measure of functional mobility and fall risk in older adults. Participants were instructed to walk at their usual pace, and the time (s) was recorded. Slower gait speed is associated with higher fall risk, reduced mobility, and lower physical function in knee osteoarthritis patients

CONTACTS AND LOCATIONS:
Overall Officials: Sema Aktürk, MD Professor, Study Chair — Inonu University
Locations (1):
- Kocaeli Health and Technology University, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
PERSONAL DATA OF PARTICIPANTS MAY BE PROVIDED TO A REASONABLE EXTENT.